CLINICAL TRIAL: NCT02415868
Title: Development of an Ex-vivo High-throughput Screening Assay for the Vaginal Microbiota of Post-menopausal Women
Brief Title: Ex Vivo High-Throughput Assay for Vaginal Community Post-menopausal Women
Acronym: FLORA
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Collaborators: NIZO Food Research (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 500-14-0004
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Postmenopausal Syndrome
Keywords: Vaginal Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiota from Vaginal Swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low pH: Post Menopausal women with vaginal pH of 4.5 or below
- High pH: Post Menopausal women with vaginal pH of 5.5 or above

SUMMARY:
This purpose of this study is to collect vaginal microbial samples of postmenopausal women to assess the optimal conditions for cultivation and storage of the vaginal microbiota. These samples will subsequently be used to develop a high-throughput assay that mimicks the vaginal microbial community of postmenopausal women. This assay will be used to select and screen compounds that can affect the vaginal microbiota and subsequently affect related symptoms such as vaginal dryness.

DETAILED DESCRIPTION:
Vaginal swabs will be collected from post-menopausal women (5 women vaginal pH ≤4.5 and 5 women with vaginal pH≥5.5), aged 45 - 75, with at least 12 months of amenorrhea. Enough women will be screened to ensure five women for each pH range.

Using a speculum, the mid lateral vaginal wall is made visible, samples will be collected by the physician or nurse using a flocked swab. After collection, vaginal swabs will be stored immediately in adequate liquid medium at 4ºC and will be transported to the lab within 7 hours after sampling for further storage and culture of the material.

The vaginal microbiota of post-menopausal women with a vaginal pH of ≤ 4.5 and ≥ 5.5 will be characterized and compared using 16S ribosomal ribonucleic acid (rRNA) sequencing. In additional, optimal conditions for cultivation and storage of the vaginal microbiota will be examined for use in assays mimicking the vaginal microbial community of postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to study design (signed informed consent)
2. Post-menopausal women
3. Vaginal pH ≤4.5 or pH ≥5.5
4. At least 12 months of amenorrhea
5. Age ≥45 and ≤75
6. Currently in a mutually monogamous sexual relationship or not sexually active;
7. Sexually abstinent 48 hours prior to visit.
8. Willing and capable of following all study instructions; and
9. Good general health.

Exclusion Criteria:

1. Vaginal pH between >4.5 and <5.5
2. Use of topical estrogen containing product 1 week prior to enrollment
3. Use of vaginal lubricants, douches, or any products applied vaginally during the week prior to the first visit
4. Use of systemic estrogen therapy or products 6 months prior to inclusion
5. Use of a vaginal pessary during the week prior to the visit
6. Excessive alcohol usage (>4 consumptions/day or >20 consumptions/week)
7. Drug usage within past 2 years
8. A history or currently undergoing immunosuppressive drug therapy, chemotherapy, or radiation therapy
9. A medical condition which might compromise immune system functions (such as cancer, leucopenia, HIV-positive, or organ transplant)
10. Antibiotics and/or anti-fungal medication use within the last four (4) weeks
11. Induced menopause due to surgical or medical interventions, such as bilateral oophorectomy, hysterectomy, chemotherapy or radiation treatment
12. Currently diagnosed with or being treated for a genital infection or urinary tract infection, subjects who had any vaginal infection one month prior to the screening will be excluded
13. Individuals with a sexually transmitted disease (self-reported or detected by the Principal Investigator)
14. At enrollment, have any social or medical condition, or psychiatric illness that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
15. Participation in a clinical trial involving an investigational product/device within the past three months; subjects who are scheduled to participate in another clinical study concurrently.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Characterization of the microbiota | 0 hours
  By 16s rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Klinkert, MD, Principal Investigator — Department of Gynaecology, University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaban B, Links MG, Jayaprakash TP, Wagner EC, Bourque DK, Lohn Z, Albert AY, van Schalkwyk J, Reid G, Hemmingsen SM, Hill JE, Money DM. Characterization of the vaginal microbiota of healthy Canadian women through the menstrual cycle. Microbiome. 2014 Jul 4;2:23. doi: 10.1186/2049-2618-2-23. eCollection 2014. PMID 25053998
- [Background] Hummelen R, Macklaim JM, Bisanz JE, Hammond JA, McMillan A, Vongsa R, Koenig D, Gloor GB, Reid G. Vaginal microbiome and epithelial gene array in post-menopausal women with moderate to severe dryness. PLoS One. 2011;6(11):e26602. doi: 10.1371/journal.pone.0026602. Epub 2011 Nov 2. PMID 22073175